CLINICAL TRIAL: NCT01122953
Title: Bioequivalence Study Of 5ml Dose Of PHENYTOIN 125mg/ 5ml Suspension Made By Laboratorios Pfizer, S.A. De C.V. Versus EPAMIN® 125 mg/5ml Made By McNeil LA LLC, Study In Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study Of PHENYTOIN Suspension Made By Pfizer, Versus EPAMIN® Made By McNeil LA LLC In Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A4121009
Record Dates: First submitted 2010-04-29; First posted 2010-05-13 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Bioequivalence; EPAMIN; PHENYTOIN
MeSH Terms: interventions — Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenytoin (Experimental)
  Interventions: Drug: Phenytoin
- Epamin (Active Comparator)
  Interventions: Drug: Epamin

INTERVENTIONS:
Drug: Phenytoin — Single dose of Phenytoin 125 mg/5 ml suspension made by Laboratorios Pfizer, S.A. de C.V.
  Arms: Phenytoin
Drug: Epamin — Single dose Epamin 125 mg/5 ml suspension made by McNeil LA LLC
  Arms: Epamin

SUMMARY:
To investigate the bioequivalence between two compounds (phenytoin and epamin) by a randomized, single dose study under fasting conditions in healthy volunteers.

DETAILED DESCRIPTION:
Bioequivalence study in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 18 to 26.9 kg/m2 or ± 10% variation of the ideal weight; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC): The AUC from administration to the last sampling time will be determined by the trapezoid method. | 0-168 h
Maximum Concentration (Cmax): The maximum plasmatic concentration (Cmax) will be obtained as the highest concentration observed in the sampling interval. | 0-168 h
Time maximum concentration (tmax) is observed. Will be reported as the time at which the maximum concentration is observed. | 0-168 h

SECONDARY OUTCOMES:
Constant of elimination (ke): Will be determined as the slope from the linear logarithmic regression of the terminal phase of the logarithmic graph of concentration over time. | 0-168 h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Mexico City, Mexico City, Mexico